CLINICAL TRIAL: NCT05418075
Title: Evaluation of the Effectiveness of Add-on Hometreatment to Family Based Therapy in Adolescent Anorexia Nervosa. A Randomised Controlled Clinical Trial
Brief Title: Evaluation of the Effectiveness of Add-on Hometreatment to Family Based Therapy in Adolescent Anorexia Nervosa.
Acronym: HTED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTED 2021-01706
Record Dates: First submitted 2022-01-05; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Anorexia in Adolescence
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Treatment as add on to Familiy-based Treatment (Experimental)
  Interventions: Other: Psychotherapy
- Familiy-based Treatment (Active Comparator)
  Interventions: Other: Psychotherapy
- Mindfulness based stress reduction training (Active Comparator)
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — If the families agree to participate in the study, they are randomly assigned to a treatment group. In each of the three groups, they are treated with FBT in a weekly session. In the two comparison groups, Hometreatment or MBSR are offered in addition to FBT, with two consultations per week in each case.

SUMMARY:
The project serves to evaluate a new treatment method with outreach services as a supplement to family-based therapy in the treatment of children and adolescents with eating disorders.

The project is intended to help identify different family structures and which families will benefit most from the new outreach service of home-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 12 -20 years.
* Successful registrations in the special consultation for eating disorders at the Clinic for Child and Adolescent Psychiatry and Psychotherapy (KJPP) of the Psychiatric University Hospital (PUK) Zurich.
* Diagnosis of anorexia nervosa or atypical anorexia nervosa (ICD-10 F50.00/ F50.01/ F50.1)
* Existing informed consent of patients* (14 years and older) and parents or legal guardians (12-14 years).
* IQ over 75
* Resident in the canton of Zurich
* Good knowledge of German

Exclusion Criteria:

* No written consent
* Children under 12 years
* Other forms of eating disorders apart from anorexia nervosa or atypical anorexia nervosa.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptomatic improvement | 3 months
  Change of the reported BMI; Weight in Kg and Height in cm will be combined to report BMI in kg/m^2
Symptomatic improvement | 3 months
  Change of the Eating Disorder Examination Interview (EDE) total score analyze using a linear random coefficient regressions model
Symptomatic improvement | 3 months
  Change of the Eating Disorder Inventory (EDI) total score analyze using a linear random coefficient regressions model

SECONDARY OUTCOMES:
State of health improvement | 3 months
  Change of the Perceived stress scale (PSS) total score measering level of perceived stress and change of the total score in Brief dyadic scale of expressed emotion (BDSEE) measering level of expressed emotion.
Remission rate | 12 months
  Remission is definde as a Body weight within 15% deviation of the normal weight and clinically unremarkable values in the EDE and EDI

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Universitätsklilnik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Besse-Flutsch N, Buhlmann C, Fabijani N, Ruschetti GG, Smigielski L, Pauli D. Home treatment as an add-on to family-based treatment for adolescents with anorexia nervosa compared with standard family-based treatment and home-based stress reduction training: study protocol for a randomized clinical trial. J Eat Disord. 2023 Aug 14;11(1):135. doi: 10.1186/s40337-023-00861-5. PMID 37580810